CLINICAL TRIAL: NCT00639600
Title: Transplantation d'îlots pancréatiques allogéniques Adultes Pour le Traitement du diabète insulinodépendant. Etude GRAGIL 1
Brief Title: Transplantation of Pancreatic Islets in Patients With Type 1 Diabetes Mellitus and Functional Kidney Graft
Acronym: GRAGIL1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: a new study has began recently
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Pierre-Yves Benhamou, University Hospital, Grenoble
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95/CHUG/10/C2
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: human pancreatic islet transplantation — human pancreatic islet transplantation

SUMMARY:
This research project is supported by a multicentric network of collaborators whose goal is to assess the efficacy of transplanting allogenic pancreas islets to restore insulin secretion in patients with type 1, insulin-dependent diabetes mellitus with kidney transplantation and to improve their metabolic control.

DETAILED DESCRIPTION:
The main objective is to demonstrate the beneficial effect of islet allotransplantation in patients with type 1 diabetes with no endogenous insulin secretion, and with a functional kidney graft. The other objectives are to evaluate the conditions for the efficacy of islet cell transplantation, to assess the improvement in quality of life and the cost of the islet cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Disease duration > 5 years
* ketose antecedents
* Basal and stimulated plasma C-< 0.2 ng/ml,<0.06 nmol/l (glycemia must be measured simultaneously_ 1.20 g/l or 6.6 mM, stimulation with glucagon IV 1 mg -Measured at à T0 and T 6 min)
* Established kidney graft ≥ 6 months
* Current creatinine clearance: ≥ 50 ml/min/1.73 m² and Proteinuria < 0.5 g/24h
* HbA1C< 12%

Exclusion Criteria:

* Hemostasis problems
* Documented hepatic pathology
* Patient under 18 or over 65 year-old
* Women with body weight over 70 kg (tolerance of 2 kg between inclusion day and transplantation day) or BMI > 26
* Men with body weight > 75 kg (tolerance of 3 kg between inclusion day and transplantation day) or BMI > 26
* insuline needs > 0.7 U/kg/j or 50 U/j
* Serious life-threatening pathology
* untreated hyperlipidemia
* Hypersensitivity to drugs rapamycine-alike
* Liver disease (transaminases or total bilirubin ≥ 3N)
* Failure to communicate or cooperate with the investigator

Exclusion criteria that are specific to the use of Rapamycine

* Hypercholesterolemia (> 350mg/dl, 9,1 mmol/l) not controlled
* Hypertriglyceridemia (> 500 mg/dl, 5,6 mmol/l) not controlled
* Leukocytes > 4500 /mm3 , neutrophils > 2000/ mm3, platelets > 100000/ mm3
* Any clinical or biological pathology that could interfere with the study
* Past or present neoplasia (with the exception of non melanoma skin cancers)
* Any hemostasis disorder needing a prolonged treatment with anticoagulation drugs. Low-dose aspirin is permitted.
* Pregnancy, lactation, pregnancy project or absence of efficient contraception
* Any medical or psychosocial condition susceptible to interfere with the study, such as drug abuse or recent alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rate of insulin-independence at 6 and 12 months after transplantation, duration of insulin-independence, survival curves | 12 months

SECONDARY OUTCOMES:
Tolerance (Measurement of portal pressure during islet injection) Quality of life (Questionnaires SF-36 and DQOL at inclusion time, then every 6 months during their waiting period and then 6 months and 12 months after transplantation) Costs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Y Benhamou, MD, PhD, Principal Investigator — University Hospital of Grenoble, Department of Endocrinology
Locations (7):
- France (6):
  - University Hospital, Besançon
  - University Hospital, Department of Endocrinology, Grenoble
  - University Hospital, Department of Endocrinology, Lyon
  - University Hospital, Department of Endocrinology, Montpellier
  - University Hospital, Department of Endocrinology, Nancy
  - University Hospital, Department of Endocrinology, Strasbourg
- University Hospital, Department of Surgery, Geneva, Switzerland

REFERENCES:
- [Derived] Lablanche S, Borot S, Wojtusciszyn A, Bayle F, Tetaz R, Badet L, Thivolet C, Morelon E, Frimat L, Penfornis A, Kessler L, Brault C, Colin C, Tauveron I, Bosco D, Berney T, Benhamou PY; GRAGIL Network. Five-Year Metabolic, Functional, and Safety Results of Patients With Type 1 Diabetes Transplanted With Allogenic Islets Within the Swiss-French GRAGIL Network. Diabetes Care. 2015 Sep;38(9):1714-22. doi: 10.2337/dc15-0094. Epub 2015 Jun 11. PMID 26068866